CLINICAL TRIAL: NCT05667961
Title: Predictors of Functional Remission in Discharged Patients With Schizophrenia After Long-term Drug Discontinuation: a Case-control Study
Brief Title: Predictors of Functional Remission in Discharged Patients With Schizophrenia After Long-term Drug Discontinuation
Status: Completed | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-TX-007
Record Dates: First submitted 2022-09-06; First posted 2022-12-29 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- the function remitted off-medicine group: * Off-medicine definition: Continuous antipsychotic maintenance therapy for at least two years before drug discontinuation and drug discontinuation of all reasons (treatment benefits, adverse events, socioeconomic difficulties, migration, stigma, etc.) for at least one year;
  * Function remitted definition: Meet the criteria of functional remission in both WHOQoL-BREF (overall points ≥ 60) and FROGS (social functioning dimension points ≥ 33, daily life dimension points ≥ 12, and treatment dimension points ≥ 12)
- the function not-remitted off-medicine group: * Off-medicine definition: Continuous antipsychotic maintenance therapy for at least two years before drug discontinuation and drug discontinuation of all reasons (treatment benefits, adverse events, socioeconomic difficulties, migration, stigma, etc.) for at least one year;
  * Function not-remitted definition: Fail to meet the criteria of functional remission in both WHOQoL-BREF and FROGS
- the function remitted on-medicine group: * On-medicine definition: Continuous antipsychotic maintenance therapy during the time this study is conducted
  * Function remitted definition: Meet the criteria of functional remission in both WHOQoL-BREF and FROGS
- the function not-remitted on-medicine group: * On-medicine definition: Continuous antipsychotic maintenance therapy during the time this study is conducted
  * Function not-remitted definition: Fail to meet the criteria of functional remission in both WHOQoL-BREF and FROGS

SUMMARY:
Study objectives:

1. Describe the characteristics of discharged patients with schizophrenia achieving functional remission after drug discontinuation.
2. Establish a prediction model of patients with schizophrenia having good prognosis after drug discontinuation.

DETAILED DESCRIPTION:
There are 2 clinically important and urgent questions to be explored in this study: 1. Who is more likely to benefit from guided drug reduction or discontinuation? How to design an individualized treatment plan which can balance the risk of relapse and side-effects from antipsychotics? 2. What are the predictors of functional remission in patients with schizophrenia after drug discontinuation? This will be the first related study to be conducted in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the diagnostic criteria of the International Classification of diseases, 10th edition (ICD-10) for a diagnosis of schizophrenia;
* Aged between 18 to 65 years old at time of investigation;
* Hospitalized in Shanghai Mental Health Center any time from the year 2013 to 2018;
* Informed consent.

Exclusion Criteria:

* Patients with neurological diseases, severe somatic diseases, psychoactive substance abuse, mental retardation, agitation, stupor, or risk of suicide, and female patients who are pregnant or breast-feeding, will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited from Shanghai Mental Health Center (SMHC), Shanghai, China
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Functional remission dimension 1 | Up to 28 weeks
  World Health Organization Quality of Life abbreviated version（WHOQoL-BREF), score from 26 to 130. Higher score indicates better functional remission.
Functional remission dimension 2 | Up to 28 weeks
  Functional Remission of General Schizophrenia Scale (FROGS), scale from 19 to 95. Higher score indicates better functional remission.

SECONDARY OUTCOMES:
Symptom assessment dimension 1 | Up to 28 weeks
  the Positive and Negative Syndrome Scale (PANSS), score from 30 to 210. High score indicates severe symptoms.
Symptom assessment dimension 2 | Up to 28 weeks
  Clinical Global Impression (CGI), score from 1 to 7. High score indicates severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Dengtang Liu, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be securely protected and will not be shared to other researchers.

REFERENCES:
- [Background] Fitzgerald P, de Castella A, Arya D, Simons WR, Eggleston A, Meere S, Kulkarni J. The cost of relapse in schizophrenia and schizoaffective disorder. Australas Psychiatry. 2009 Aug;17(4):265-72. doi: 10.1080/10398560903002998. PMID 19585288
- [Background] Kane JM. Treatment strategies to prevent relapse and encourage remission. J Clin Psychiatry. 2007;68 Suppl 14:27-30. PMID 18284275
- [Background] Takeuchi H, Siu C, Remington G, Fervaha G, Zipursky RB, Foussias G, Agid O. Does relapse contribute to treatment resistance? Antipsychotic response in first- vs. second-episode schizophrenia. Neuropsychopharmacology. 2019 May;44(6):1036-1042. doi: 10.1038/s41386-018-0278-3. Epub 2018 Nov 22. PMID 30514883
- [Background] De Hert M, Sermon J, Geerts P, Vansteelandt K, Peuskens J, Detraux J. The Use of Continuous Treatment Versus Placebo or Intermittent Treatment Strategies in Stabilized Patients with Schizophrenia: A Systematic Review and Meta-Analysis of Randomized Controlled Trials with First- and Second-Generation Antipsychotics. CNS Drugs. 2015 Aug;29(8):637-58. doi: 10.1007/s40263-015-0269-4. PMID 26293744
- [Background] Sampson S, Joshi K, Mansour M, Adams CE. Intermittent drug techniques for schizophrenia. Schizophr Bull. 2013 Sep;39(5):960-1. doi: 10.1093/schbul/sbt096. Epub 2013 Jul 16. PMID 23861538
- [Background] Tiihonen J, Tanskanen A, Taipale H. 20-Year Nationwide Follow-Up Study on Discontinuation of Antipsychotic Treatment in First-Episode Schizophrenia. Am J Psychiatry. 2018 Aug 1;175(8):765-773. doi: 10.1176/appi.ajp.2018.17091001. Epub 2018 Apr 6. PMID 29621900
- [Background] Gaebel W, Stricker J, Riesbeck M. The long-term antipsychotic treatment of schizophrenia: A selective review of clinical guidelines and clinical case examples. Schizophr Res. 2020 Nov;225:4-14. doi: 10.1016/j.schres.2019.10.049. Epub 2019 Dec 2. PMID 31806527
- [Background] Zito MF, Marder SR. Rethinking the risks and benefits of long-term maintenance in schizophrenia. Schizophr Res. 2020 Nov;225:77-81. doi: 10.1016/j.schres.2019.10.057. Epub 2019 Dec 2. PMID 31806525
- [Background] Haijma SV, Van Haren N, Cahn W, Koolschijn PC, Hulshoff Pol HE, Kahn RS. Brain volumes in schizophrenia: a meta-analysis in over 18 000 subjects. Schizophr Bull. 2013 Sep;39(5):1129-38. doi: 10.1093/schbul/sbs118. Epub 2012 Oct 5. PMID 23042112
- [Background] Morgan C, Lappin J, Heslin M, Donoghue K, Lomas B, Reininghaus U, Onyejiaka A, Croudace T, Jones PB, Murray RM, Fearon P, Doody GA, Dazzan P. Reappraising the long-term course and outcome of psychotic disorders: the AESOP-10 study. Psychol Med. 2014 Oct;44(13):2713-26. doi: 10.1017/S0033291714000282. Epub 2014 Feb 26. PMID 25066181
- [Background] Wunderink L, Nienhuis FJ, Sytema S, Slooff CJ, Knegtering R, Wiersma D. Guided discontinuation versus maintenance treatment in remitted first-episode psychosis: relapse rates and functional outcome. J Clin Psychiatry. 2007 May;68(5):654-61. doi: 10.4088/jcp.v68n0502. PMID 17503973
- [Background] Wils RS, Gotfredsen DR, Hjorthoj C, Austin SF, Albert N, Secher RG, Thorup AA, Mors O, Nordentoft M. Antipsychotic medication and remission of psychotic symptoms 10years after a first-episode psychosis. Schizophr Res. 2017 Apr;182:42-48. doi: 10.1016/j.schres.2016.10.030. Epub 2016 Oct 27. PMID 28277310
- [Background] Hui CLM, Honer WG, Lee EHM, Chang WC, Chan SKW, Chen ESM, Pang EPF, Lui SSY, Chung DWS, Yeung WS, Ng RMK, Lo WTL, Jones PB, Sham P, Chen EYH. Long-term effects of discontinuation from antipsychotic maintenance following first-episode schizophrenia and related disorders: a 10 year follow-up of a randomised, double-blind trial. Lancet Psychiatry. 2018 May;5(5):432-442. doi: 10.1016/S2215-0366(18)30090-7. Epub 2018 Mar 15. PMID 29551618
- [Background] Boyer L, Richieri R, Guedj E, Faget-Agius C, Loundou A, Llorca PM, Auquier P, Lancon C. Validation of a functional remission threshold for the Functional Remission of General Schizophrenia (FROGS) scale. Compr Psychiatry. 2013 Oct;54(7):1016-22. doi: 10.1016/j.comppsych.2013.04.008. Epub 2013 May 31. PMID 23731897
- [Background] Silva SM, Santana ANC, Silva NNBD, Novaes MRCG. VES-13 and WHOQOL-bref cutoff points to detect quality of life in older adults in primary health care. Rev Saude Publica. 2019 Apr 1;53:26. doi: 10.11606/S1518-8787.2019053000802. PMID 30942268
- [Background] Gorwood P, Mallet J, Lancrenon S. Functional remission in schizophrenia: A FROGS-based definition and its convergent validity. Psychiatry Res. 2018 Oct;268:94-101. doi: 10.1016/j.psychres.2018.07.001. Epub 2018 Jul 3. PMID 30015112
- [Background] Matza LS, Phillips GA, Revicki DA, Ascher-Svanum H, Malley KG, Palsgrove AC, Faries DE, Stauffer V, Kinon BJ, Awad AG, Keefe RS, Naber D. Validation of a patient interview for assessing reasons for antipsychotic discontinuation and continuation. Patient Prefer Adherence. 2012;6:521-32. doi: 10.2147/PPA.S25635. Epub 2012 Jul 13. PMID 22879738
- [Background] Matza LS, Phillips GA, Revicki DA, Ascher-Svanum H, Kaiser D, Stauffer V, Shorr JM, Kinon BJ. Development of a clinician questionnaire and patient interview to assess reasons for antipsychotic discontinuation. Psychiatry Res. 2011 Oct 30;189(3):463-8. doi: 10.1016/j.psychres.2011.05.030. Epub 2011 Jun 17. PMID 21684017
- [Background] Matza LS, Phillips GA, Revicki DA, Ascher-Svanum H, Malley KG, Palsgrove AC, Faries DE, Stauffer V, Kinon BJ, George Awad A, Keefe RS, Naber D. Validation of a clinician questionnaire to assess reasons for antipsychotic discontinuation and continuation among patients with schizophrenia. Psychiatry Res. 2012 Dec 30;200(2-3):835-42. doi: 10.1016/j.psychres.2012.05.005. Epub 2012 Jul 28. PMID 22841345
- [Derived] Lu C, Dong Y, Zhai Z, Gao T, Luo M, Feng T, Ma X, Chang D, Chen J, Xue J, Zhao Y, Li X, Shao C, Liu D. Prediction of functional remission in patients with schizophrenia after antipsychotic discontinuation (FURSAD): protocol for a real-world case-control study. BMJ Open. 2024 Dec 27;14(12):e087645. doi: 10.1136/bmjopen-2024-087645. PMID 39732483